CLINICAL TRIAL: NCT03915392
Title: Diffusion Weighted MRI Accuracy in Cholesteatoma Localization
Acronym: CHOLEMRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7122
Record Dates: First submitted 2018-09-14; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2018-09

CONDITIONS: Cholesteatoma
Keywords: Diffusion weighted MRI; Cholesteatoma; Localization
MeSH Terms: conditions — Cholesteatoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Magnetic resonance imaging of the middle ear has an increasing place in the therapeutic strategy in otology and especially for cholesteatoma. It is currently performed for complicated cholesteatomas and as part of the follow-up of operated patients to detect a recurrence or a cholesteatoma residue (alternative of choice to "second look" surgery). Some people take CT and MRI fusion to improve the localization of cholesteatoma. Many studies have investigated the diagnostic capabilities of MRI but very few have demonstrate their reliability in location diagnosis. The aim of the study was to propose a topographic reading method of the MRI of the middle ear and to evaluate the performances in the localization of the cholesteatoma in order to adapt the surgical management

ELIGIBILITY:
inclusion criteria

* Age: from 1 month and up
* Sex: man / woman
* Patient who had a tympanoplasty in closed technique, for the first surgical time of a cholesteatoma or for residual or recurrent cholesteatoma, performed by the same radiologist (Pr Anne Charpiot) with the following characteristics:

  * Code of the Common Classification of Medical Acts (CCAM)

    * Exeresis of cholesteatoma with tympanoplasty in closed technique and ossiculoplasty (CBFA002)
    * Exeresis of cholesteatoma with tympanoplasty in closed technique (CBFA006)
    * Exeresis of cholesteatoma confined to the tympanic cavity without antro-attic exploration (CBFA005)
    * Tympanoplasty in closed technique with posterior tympanotomy (CBMD001)
    * Secondary tympanoplasty in closed technique (CBMD002)
  * Diagnostic code of the International Classification of Diseases (ICD10)

    * Cholesteatoma of the middle ear (H71)
* Diagnosis of macroscopic and / or pathological cholesteatoma.
* Preoperative diagnosis of cholesteatoma on MRI of the middle ear performed in less than 6 months by the same radiologist (Pr Francis Veillon).
* Subject (or the holders of parental authority in the case of minors) having agreed to the use of medical data for the purpose of this research.

Cholesteatoma is a very common disease in the pediatric population, with important functional issues, whose treatment is surgical. That's why our study includes minor subjects.

Criteria of non-inclusion

* Refusal of the patient to participate in the study
* Absence of data concerning the diagnosis and / or localization of cholesteatoma on the operative record
* Subject under the protection of justice
* Subject under guardianship or curatorship
* Pregnancy (woman of childbearing age)
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent cholesteatoma surgery between January 1, 2010 and December 31, 2017
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
MRI imaging study to locate cholesteatoma. | The period from January 1st, 2010 to Dcember 31, 2017 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Anne CHARPIOT, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service D'Orl Et de Chirurgie Cervico-Faciale, Strasbourg, France